CLINICAL TRIAL: NCT02027363
Title: Maintenance Treatment With Capecitabine Versus Observation After First Line Chemotherapy in Patients With Metastatic Colorectal Cancer: a Randomized Phase II Study
Brief Title: Maintenance Treatment With Capecitabine in Colorectal Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ruihua Xu, Sun Yat-sen University cancer center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Maintenance study
Record Dates: First submitted 2013-12-15; First posted 2014-01-06 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2014-01

CONDITIONS: Colorectal Neoplasms; Neoplasms Metastasis
Keywords: Metastasis colorectal cancer; Maintenance; First-line treatment; Capecitabine
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Capecitabine; Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Observation group (Experimental): Patients with metastatic colorectal cancer who achieved objective response or stable disease after 4-6 months first-line chemotherapy would stop the chemotherapy and observation.
  Interventions: Other: Observation
- Capecitabine group (Experimental): Patients with metastatic colorectal cancer who achieved objective response or stable disease after 4-6 months first-line chemotherapy could continue to receive oral capecitabine as maintenance therapy, capecitabine, 1000mg/m2 bid d1-14, every 3 week.
  The maintenance treatment was continued until progression, unacceptable toxicity, or patient withdrawal.
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Capecitabine — maintenance with apecitabine，1,000 mg/m2 twice a day， days1-15，every 3 weeks，until progression, unacceptable toxicity, or patient withdrawal.
  Other Names: Capecitabine (XELODA ，Roche)
  Arms: Capecitabine group
Other: Observation — Patients with metastatic colorectal cancer who achieved objective response or stable disease after 4-6 months first-line chemotherapy would stop the chemotherapy and observation
  Arms: Observation group

SUMMARY:
Colorectal cancer is one of the most common malignant tumors, with the morbidity of approximate 100 million cases per year. About 40% of patients present with metastatic (stage IV) colorectal cancer at the time of diagnosis, and about 25% of patients with local lesion will ultimately develop metastatic disease.

5-Fluorouracil（5-FU) was the only efficacious treatment for metastatic colorectal cancer before the nineties of the 20th century, and afterwards as the discovery of chemotherapy such as oxaliplatin, irinotecan and capecitabine, response rate as well as survival had been improved greatly.

Most of advanced colorectal cancer will progress after first-line treatment; therefore, seeking an efficient and low toxic maintaining regimen to prolong PFS becomes a hot topic in oncologic field. Some clinical researches demonstrated that maintaining treatment followed first-line treating advanced NSCLC could extend PFS and OS. In metastatic colorectal cancer, patients receiving 5-FU/leucovorin(LV) maintaining therapy experienced significantly longer PFS than that stopped chemotherapy after six cycles of FOLFOX4 in OPTIMOX2 study. One phase II study shown that median PFS was 13.9 months, and median OS was 31 months in 30 patients receiving first-line treatment of six- month FOLFOX4 followed by UFT as maintaining treatment . A non-randomized small sample study conducted in department of medical oncology of Sun Yat-Sen University Cancer Center indicated that patients receiving first-line treatment of XELOX followed by capecitabine as maintaining therapy has significantly prolonged median TTP, comparing with the non-maintaining treatment patients,(14months vs. 9 month, respectively).

Above all, so far, there is no data to demonstrate that regular 4-6 month chemotherapy followed by maintaining treatment could prolong TTP and OS for advanced colorectal cancer. Capecitabine is effective for colorectal cancer, and was approved as palliative treatment for advanced colorectal cancer and adjuvant chemotherapy; in addition, with its relative less frequency of side effects and convenient oral administration, capecitabine as maintaining regimen could be prone to be accepted by patients. Therefore, our study is designed to investigate that capecitabine as maintaining treatment after first-line palliative chemotherapy could improve TTP and OS for patients with advanced colorectal cancer through a perspective randomized clinical study.

DETAILED DESCRIPTION:
Patients with metastatic colorectal cancer who achieved objective response or stable disease after 4-6 months first-line chemotherapy were randomly assigned to one of two groups, to receive either capecitabine (2000 mg/m2 per day on days 1-14,Q3W) as maintenance therapy or observation. The treatment will continue until disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* age older than 18 years
* Eastern Cooperative Oncology Group performance status (ECOG PS) 0-1
* histologically confirmed colorectal cancer with inoperable locally advanced or recurrent and/or metastatic disease, not amenable to curative therapy.
* Life expectancy of at least 3 months
* Hematologic, Biochemical and Organ Function 14. Neutrophil count < 1.5 × 109/L, or platelet count < 100 × 109/L. 15. Serum bilirubin > 1.5 × upper limit of normal (ULN); or, AST or ALT > 2.5 × ULN (or > 5 × ULN in patients with liver metastases); or, alkaline phosphatase > 2.5 × ULN (or > 5 × ULN in patients with liver metastases, or > 10 × ULN in patients with bone but no liver metastases); or albumin < 25 g/L
* Patients who achieved objective response or stable disease after 16-24 weeks first line chemotherapy
* Signed informed consent

Exclusion Criteria:

* Known hypersensitivity to capecitabine
* History or clinical evidence of brain metastases
* No previous chemotherapy for metastatic disease
* Positive serum pregnancy test in women of childbearing potential
* Subjects with reproductive potential not willing to use an effective method of contraception
* Received any investigational drug treatment within 4 weeks of start of study treatment
* other prior malignancies in the past 5 years
* unresolved bowel obstruction or malabsorption syndrome

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Estimated)
Dates: Start 2010-01; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
progression-free survival (PFS) | up to 30 months
  defined as the interval between initial treatment and the first documentation of disease progression or death

SECONDARY OUTCOMES:
overall survival (OS) | up to 3 years
  measured from the initiation of chemotherapy to the date of the last follow-up or death
overall response(ORR) | up to 9 months
  Overall tumor response: This is defined as the occurrence of either a confirmed complete (CR) or a partial (PR) best overall response as determined by the RECIST criteria from confirmed radiographic evaluations of target and non-target lesions.
Safety | 3 years
  Adverse events and laboratory tests graded according to the NCI-CTC AE Version 4.

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Xu, M.D,Ph.D, Principal Investigator — Sun Yat-sen University
Locations (1):
- Medical Oncology,Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Result] Li YH, Luo HY, Wang FH, Wang ZQ, Qiu MZ, Shi YX, Xiang XJ, Chen XQ, He YJ, Xu RH. Phase II study of capecitabine plus oxaliplatin (XELOX) as first-line treatment and followed by maintenance of capecitabine in patients with metastatic colorectal cancer. J Cancer Res Clin Oncol. 2010 Apr;136(4):503-10. doi: 10.1007/s00432-009-0682-5. Epub 2009 Sep 24. PMID 19777259
- [Result] Waddell T, Gollins S, Soe W, Valle J, Allen J, Bentley D, Morris J, Lloyd A, Swindell R, Taylor MB, Saunders MP. Phase II study of short-course capecitabine plus oxaliplatin (XELOX) followed by maintenance capecitabine in advanced colorectal cancer: XelQuali study. Cancer Chemother Pharmacol. 2011 May;67(5):1111-7. doi: 10.1007/s00280-010-1322-0. Epub 2010 Jul 30. PMID 20676676
- [Derived] Luo HY, Li YH, Wang W, Wang ZQ, Yuan X, Ma D, Wang FH, Zhang DS, Lin DR, Lin YC, Jia J, Hu XH, Peng JW, Xu RH. Single-agent capecitabine as maintenance therapy after induction of XELOX (or FOLFOX) in first-line treatment of metastatic colorectal cancer: randomized clinical trial of efficacy and safety. Ann Oncol. 2016 Jun;27(6):1074-1081. doi: 10.1093/annonc/mdw101. Epub 2016 Mar 2. PMID 26940686